CLINICAL TRIAL: NCT00141323
Title: PEARL: Postmenopausal Evaluation And Risk-Reduction With Lasofoxifene
Brief Title: Postmenopausal Evaluation and Risk-reduction With Lasofoxifene (PEARL)
Acronym: PEARL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A2181002
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Lasofoxifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lasofoxifene 0.5 mg/day (Experimental)
  Interventions: Drug: lasofoxifene
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- lasofoxifene 0.25 mg/day (Experimental)
  Interventions: Drug: lasofoxifene

INTERVENTIONS:
Drug: lasofoxifene — 0.5 mg once per day, orally
  Arms: lasofoxifene 0.5 mg/day
Other: placebo — placebo
  Arms: placebo
Drug: lasofoxifene — 0.25 mg once per day, orally
  Arms: lasofoxifene 0.25 mg/day

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of 2 doses of the investigational drug, lasofoxifene, compared to placebo (an inactive substance) in reducing new spinal fractures in women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal at least 5 years; Screening bone mineral density more than or equal to 2.5 S.D.s below the mean for young adults at the lumbar spine or femoral neck.

Exclusion Criteria:

Metabolic bone disease other than osteoporosis; Taking approved medications for osteoporosis; Have had a recent osteoporotic fracture (within 1 year) and/or have a bone mineral density more than 4.5 S.D.s below the mean for young adults at the lumbar spine or femoral neck.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8556 (Estimated)
Dates: Start 2001-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
New morphometric vertebral fractures | 3 years
New cases of breast cancer | 5 years
New non-vertebral fractures | 5 years

SECONDARY OUTCOMES:
All clinical fractures, non-vertebral fractures, BMD, breast cancer, cardiovascular events, and gynecological safety events | 3 years
All clinical fractures, new morphometric vertebral fractures, BMD, cardiovascular events, and gynecological safety events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (137):
- United States (32):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Palm Desert, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Montgomery Village, Maryland
  - Pfizer Investigational Site, Arden Hills, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Centerville, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Charleroia, Pennsylvania
  - Pfizer Investigational Site, Monessen, Pennsylvania
  - Pfizer Investigational Site, Cordova, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Redmond, Washington
  - Pfizer Investigational Site, Seattle, Washington
- Argentina (6):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Capital Federal - Buenos Aires
  - Pfizer Investigational Site, Capital Federal
  - Pfizer Investigational Site, S2000dhl- Rosario - Santa Fe
- Australia (9):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Ashford, South Australia
  - Pfizer Investigational Site, Dulwich, South Australia
  - Pfizer Investigational Site, Geelong, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
  - Pfizer Investigational Site, Randwick
- Belgium (2):
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Leuven
- Brazil (2):
  - Pfizer Investigational Site, São Caetano do Sul, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Costa Rica (7):
  - Pfizer Investigational Site, Cartago, Cartago Province
  - Pfizer Investigational Site, Curridabat, Provincia de San José
  - Pfizer Investigational Site, Paseo Colon, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
  - Pfizer Investigational Site, San Pedro, Provincia de San José
  - Pfizer Investigational Site, Escazú
  - Pfizer Investigational Site, San José
- Pfizer Investigational Site, Zagreb, Croatia
- Denmark (2):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Hvidovre
- Egypt (2):
  - Pfizer Investigational Site, Cairo
  - Pfizer Investigational Site, Heliopolis, Cairo
- Estonia (3):
  - Pfizer Investigational Site, Pärnu
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Finland (3):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Turku
- France (2):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, München
- Hong Kong (2):
  - Pfizer Investigational Site, New Territories, Hong Kong
  - Pfizer Investigational Site, Shatin, New Territories
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Győr
- India (10):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Thiruvananthapuram, Kerala
  - Pfizer Investigational Site, Matunga (East), Mumbai
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Vellore, Tamil Nadu
  - Pfizer Investigational Site, Jaipur
  - Pfizer Investigational Site, New Delhi
  - Pfizer Investigational Site, Parel, Mumbai
- Ireland (2):
  - Pfizer Investigational Site, Dublin, Dublin
  - Pfizer Investigational Site, Dublin
- Italy (2):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Verona
- Japan (5):
  - Pfizer Investigational Site, 15-3-1 Maki Ohita-shi, Ohita-ken
  - Pfizer Investigational Site, Ohita, Ohita
  - Pfizer Investigational Site, 2-7-8 Yoyogi Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Tokyo
- Lithuania (3):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Vilnius
- Mexico (3):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Tlalpan, Mexico City
  - Pfizer Investigational Site, Cp 11800, Mexico Df
- Norway (4):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Hamar
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Paradis
- Poland (3):
  - Pfizer Investigational Site, Nowogrodzka 62A, Warszawa
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
- Romania (4):
  - Pfizer Investigational Site, Timișoara, Timiș County
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Iași
  - Pfizer Investigational Site, Timișoara
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- South Africa (3):
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
- Pfizer Investigational Site, Seoul, Korea, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- Pfizer Investigational Site, Gothenburg, Sweden
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Izmir
- United Kingdom (4):
  - Pfizer Investigational Site, Harrow, Middlesex
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Stanmore, Middlesex
  - Pfizer Investigational Site, Aberdeen, Scotland

REFERENCES:
- [Derived] Ensrud K, LaCroix A, Thompson JR, Thompson DD, Eastell R, Reid DM, Vukicevic S, Cauley J, Barrett-Connor E, Armstrong R, Welty F, Cummings S. Lasofoxifene and cardiovascular events in postmenopausal women with osteoporosis: Five-year results from the Postmenopausal Evaluation and Risk Reduction with Lasofoxifene (PEARL) trial. Circulation. 2010 Oct 26;122(17):1716-24. doi: 10.1161/CIRCULATIONAHA.109.924571. Epub 2010 Oct 11. PMID 20937977
- [Derived] Cummings SR, Ensrud K, Delmas PD, LaCroix AZ, Vukicevic S, Reid DM, Goldstein S, Sriram U, Lee A, Thompson J, Armstrong RA, Thompson DD, Powles T, Zanchetta J, Kendler D, Neven P, Eastell R; PEARL Study Investigators. Lasofoxifene in postmenopausal women with osteoporosis. N Engl J Med. 2010 Feb 25;362(8):686-96. doi: 10.1056/NEJMoa0808692. PMID 20181970
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2181002&StudyName=Postmenopausal%20Evaluation%20and%20Risk-reduction%20with%20Lasofoxifene%20%28PEARL%29